CLINICAL TRIAL: NCT00642187
Title: A Placebo-controlled Comparison of the Efficacy and Safety of the Current US Version of Pulmicort (Budesonide) Turbuhaler and the New Version of Pulmicort Turbuhaler in Asthmatic Adults Currently Treated With Inhaled Steroids.
Brief Title: New Version Pulmicort Turbuhaler USA Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Lars-Göran Carlsson
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SD-004-0620; D5254C00620
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma; Pulmicort; Turbuhaler; Budesonide; Flexhaler
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pulmicort
  Interventions: Drug: budesonide
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: budesonide
  Other Names: Pulmicort
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
A comparison of the safety, efficacy and budesonide pharmacokinetics of the currently approved Pulmicort Turbuhaler with a new version of the inhaler, in adult patients who have asthma and are currently being treated with inhaled steroids. In addition the study evaluated the functionality of the new inhaler at the end of its intended life.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years old with a diagnosis of asthma (as defined by the ATS) for at least 6 months.
* To enter the run in period, subjects were also required to have the following:
* A forced expiratory volume (FEV1) in 1 second of 60% to 90% of predicted normal, airway reversibility of at least 12% and 0.20 L, use of orally inhaled corticosteroids for at least 3 months prior to the study.
* At Visit 2, subjects who met additional entry criteria related to rescue medication use and asthma symptom scores during the run in period plus visit specific FEV1 requirements were assigned to randomized treatments

Exclusion Criteria:

* Life threatening asthma, Two or more overnight hospitalisations for asthma within 1 year or any emergency room visit for asthma within 6 months of starting study.
* Use of steroid tablets or injections during the month (28 days) prior to Visit 1 and use of other asthma medicines (except rescue medication) within 2 weeks prior to the study.
* Any acute exacerbation of asthma or a respiratory tract infection within 30 days prior to the study. Subject must not smoke or have smoked within 6 months of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2002-07; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Forced Expiratory Volume in 1 second | Week 2, 4 and 8, then at week 12

SECONDARY OUTCOMES:
Change from baseline in Forced Vital Capacity, Morning Peak Expiratory Flow, Daytime and nighttime asthma symptom scores, beta-agonist use and discontinuation rate. | Week 2, 4 and 8, then at week 12
Incidence of Adverse Events | Week 2,4 and 8, then at week 12
Pharmacokinetics of budesonide (AUC, maximum concentration and time to maximum concentration) | 6 or 12 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Bertil Andersson, Study Director — AZ employee; Lars-Göran Carlsson, Study Director — AZ employee